CLINICAL TRIAL: NCT01287533
Title: Efficacy of Monthly Ibandronate in Women With Rheumatoid Arthritis and Reduced Bone Mineral Density Receiving Long-term Glucocorticoids
Brief Title: Efficacy of Monthly Ibandronate in Women With RA and Reduced Bone Mineral Density Receiving Long-term Steroids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yeong-Wook Song (Other)
Responsible Party: Sponsor-Investigator, Yeong-Wook Song, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 112942
Record Dates: First submitted 2011-01-30; First posted 2011-02-01 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Rheumatoid Arthritis; Osteoporosis; Osteopenia
Keywords: Rheumatoid arthritis; Glucocorticoid induced osteoporosis; Vertebral fracture
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoporosis; Bone Diseases, Metabolic; Spinal Fractures | interventions — Ibandronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibandronate treatment (Experimental): Ibandronate 150mg PO once every 4 weeks
  Interventions: Drug: Ibandronate
- Placebo arm (Placebo Comparator): Placebo PO once every 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibandronate — monthly dosage of ibandronate 150mg
  Arms: Ibandronate treatment
Drug: Placebo — monthly dosage of placebo
  Arms: Placebo arm

SUMMARY:
This study was to investigate the efficacy of oral monthly ibandronate in the management of glucocorticoid induced osteoporosis in women with rheumatoid arthritis.

DETAILED DESCRIPTION:
Glucocorticoid therapy is associated with a number of significant side effects, of which bone loss resulting in glucocorticoid-induced osteoporosis and an increase in fracture risk is the most serious. However studies show that many patients treated with glucocorticoids do not receive treatment to prevent bone loss. There exist 5 large randomized controlled clinical trials providing evidence that the bisphosphonates etidronate, alendronate, and risedronate are effective in both the prevention and the treatment of glucocorticoid-induced osteoporosis. Significant increases in BMD with bisphosphonate treatment, most consistently observed in lumbar spine, were seen in patients with many different glucocorticoid-treated disorders; most often RA and polymyalgia rheumatica, and occurred generally irrespective of patient age, sex and menopausal status in women. In addition, statically significant reductions in the absolute risk and relative risk of incident radiographic vertebral fractures were demonstrated after 1 year of treatment with risedronate. A similar significant reduction in the risk of incident radiographic vertebral fractures was seen in alendronate treated patients who completed 2 years of a study of alendronate in the prevention and treatment of glucocorticoid-induced osteoporosis. There exists a data about Ibandronate which reported that intermittent intravenous ibandronate reduced vertebral fracture risk in corticosteroid-induced osteoporosis. However, there is no report about oral monthly ibandronate. Current oral bisphosphonates, which are given either daily or weekly, are associated with stringent, inconvenient dosing schedules. Less frequent dosing may provide great acceptability. The objective of this study was to investigate the efficacy of oral monthly ibandronate in women receiving long-term glucocorticoids.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis fulfilling the 1987 ACR criteria
* Women equal and above 18 years, less than 75 years old
* L1-4 T score less than -1.0 and equal or above -3.0 SD measured by DXA (Dual Energy X-ray Absorptiometry)
* Patient must have taken prednisolone 5mg or its equivalent for more than 3 consecutive months within 1 year
* Patient who would be taking glucocorticoids for more than 3 months after enrollment

Exclusion Criteria:

* Patient with vertebral fractures or nonvertebral fractures associated with osteoporosis
* Patient diagnosed with malignancy within 5 years
* Patient with endocrine dysfunction
* RA functional class 4
* Patient who took bisphosphonates within 6 months
* Patient on medication affecting bone mineral metabolism

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2010-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Changes in L1-4 bone mineral density compared with baseline | 48 weeks

SECONDARY OUTCOMES:
Changes in femur bone mineral density compared with baseline | 48 weeks
Changes in L1-4 and femur bone mineral density compared with baseline | 24 weeks
Changes in C-telopeptide compared with baseline | 24 and 48 weeks
Cumulative incidence of vertebral fracture | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Shin K, Park SH, Park W, Baek HJ, Lee YJ, Kang SW, Choe JY, Yoo WH, Park YB, Song JS, Lee SG, Yoo B, Yoo DH, Song YW. Monthly Oral Ibandronate Reduces Bone Loss in Korean Women With Rheumatoid Arthritis and Osteopenia Receiving Long-term Glucocorticoids: A 48-week Double-blinded Randomized Placebo-controlled Investigator-initiated Trial. Clin Ther. 2017 Feb;39(2):268-278.e2. doi: 10.1016/j.clinthera.2017.01.008. Epub 2017 Feb 1. PMID 28161119